CLINICAL TRIAL: NCT01805024
Title: Congenital Muscular Dystrophy Ascending Multiple Dose Cohort Study Analyzing Pharmacokinetics at Three Dose Levels In Children and Adolescents With Assessment of Safety and Tolerability of Omigapil (CALLISTO)
Acronym: CALLISTO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNT-I-015; FDA-OPD 5076 (Other: FDA); NCT02326831 (obsolete NCT alias)
Record Dates: First submitted 2013-03-04; First posted 2013-03-05 (Estimated); Results first posted 2019-09-20 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Congenital Muscular Dystrophy
MeSH Terms: interventions — dibenzo(b,f)oxepin-10-ylmethyl-methyl-prop-2-ynyl-amine

ARMS (1):
- Omigapil (Experimental): Omigapil treatment oral administration once per day after breakfast Cohort 1 Cohort 1 0.02 mg/kg/day Cohort 2 0.08 mg/kg/day Cohort 3a 0.04 mg/kg/day Cohort 3b 0.06 mg/kg/day
  Interventions: Drug: Omigapil

INTERVENTIONS:
Drug: Omigapil — Cohort 1 0.02 mg/kg/day Cohort 2 0.08 mg/kg/day Cohort 3a 0.04 mg/kg/day Cohort 3b 0.06 mg/kg/day

SUMMARY:
The purpose of the study is to establish the pharmacokinetic profile of omigapil in paediatric and adolescent patients with CMD and to evaluate the safety and tolerability of omigapil.

Funding source - FDA OOPD

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory and non-ambulatory patients from age 5 - 16 years (5 years old and <17 years old) at time of screening with a clinical picture (see below) consistent with COL6-related dystrophy (COL6-RD) or LAMA2-related dystrophy (LAMA2-RD)
* Under regular review at a neuromuscular center
* On adequate double-barrier contraception (if of child-bearing potential)
* Stable on any allowed concomitant medications for 1 month prior to run in Phase
* Forced Vital Capacity (FVC) 30-80% of the predicted value and confirmed at Screening and Baseline visit(s)

For patients with Collagen VI-related dystrophy (COL6-RD)- required clinical picture:

• Muscle weakness: inability to walk or, if patient is still ambulatory, inability to run and > 5 s for 10 m walk

Genetic and Pathology:

• Molecular diagnosis of COL6-RD, defined by one dominant or two recessive mutation(s) in COL6A1, COL6A2 or COL6A3 known to cause the clinical picture,,

OR

• Histological diagnosis showing (i) absent or significantly decreased expression of collagen VI in muscle (overall reduction or basal lamina specific) or (ii) absent or significantly abnormal matrix in skin fibroblast culture

For patients with Laminin alpha 2 related dystrophy (LAMA2-RD) - required clinical picture:

• Muscle weakness: Inability to walk; if patient is still ambulatory, inability to run and > 5 s for 10 m walk.

Genetics and Pathology:

• Either: 2 identified pathologic or probable pathologic mutations in LAMA2 gene

OR:

• 1 identified pathologic or probable pathologic mutation in LAMA 2 gene with evidence of decrease in laminin alpha 2 staining on muscle or skin biopsy

OR:

• Evidence of decrease in laminin alpha 2 staining on muscle or skin biopsy with matching clinical phenotype and no suspicion of alpha dystroglycanopathy (aDG-RD) (clinically or by staining on muscle biopsy)

Exclusion Criteria:

* Use of any investigational drug other than the study medication within 12 weeks of study start.
* Recurrent hospitalisation for chest infections in previous 2 years (≥2 per year)
* Patients with respiratory parameters (eg: low pulmonary function test value i.e. <30% or need for brief course of daytime non-invasive ventilation) currently affected by short term medications, or acute illness/ conditions (conduct baseline assessments when the patient has recovered and no longer taking acute medication)
* Any need for surgery (scoliosis, gastrostomy, other) in the preceding 24 weeks or foreseen during the course of the study.
* Patient has an intercurrent significant medical condition or situation which in the opinion of the Investigator or the study Medical Monitor may put the patient at significant risk, confound the study results or interfere significantly with the patient's participation in the study
* Failure to thrive, defined as:
* Falling 20 percentiles (20/100) in body weight in the 12 weeks preceding Screening/Baseline (based on family report of weight loss and acquiring relevant medical records)
* In patients below the 3rd percentile, any further drop in body weight percentile in the 12 weeks preceding Screening/Baseline (based on family report of weight loss and acquiring relevant medical records)
* Weight less than 17kg at Baseline
* Morbidly obese or grossly overweight (≥86 percentile BMI in children)
* History of epilepsy or on antiepileptic medication at Screening/Baseline
* Diabetes
* On daytime Non Invasive Ventilation (NIV)
* Intake of prohibited medication (as listed in Appendix I)
* Anticipated need for anesthesia during the course of this study
* Patients with renal impairment defined as urinary protein concentration ≥ 0.2 g/L
* Patients with moderate to severe hepatic impairment
* ALT ≥ 8x upper limit of normal (ULN) and total bilirubin 2x ULN (plus >35% 'direct' bilirubin), or
* ALT ≥ 8x ULN and INR >1.5 or ALT >2x baseline levels, and total bilirubin > 2x ULN (plus >35% 'direct' bilirubin), or
* ALT >2x baseline levels, and INR greater than 1.5,

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2014-12; Primary Completion 2017-12-05 (Actual); Study Completion 2018-01-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- NINDS, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Foley AR, Yun P, Leach ME, Neuhaus SB, Averion GV, Hu Y, Hayes LH, Donkervoort S, Jain MS, Waite M, Parks R, Bharucha-Goebel DX, Mayer OH, Zou Y, Fink M, DeCoster J, Mendoza C, Arevalo C, Hausmann R, Petraki D, Cheung K, Bonnemann CG. Phase 1 Open-Label Study of Omigapil in Patients With LAMA2- or COL6-Related Dystrophy. Neurol Genet. 2024 May 29;10(3):e200148. doi: 10.1212/NXG.0000000000200148. eCollection 2024 Jun. PMID 38915423

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 0.02 mg/kg/Day; Cohort 2 0.08 mg/kg/Day; Cohort 3a 0.04 mg/kg/Day; Cohort 3b 0.06 mg/kg/Day: Omigapil Treatment, oral administration once per day after breakfast
Period: Overall Study
Arm/Group | Cohort 1 0.02 mg/kg/Day | Cohort 2 0.08 mg/kg/Day | Cohort 3a 0.04 mg/kg/Day | Cohort 3b 0.06 mg/kg/Day
Started | 4 | 4 | 4 | 8
Completed | 4 | 4 | 4 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics per cohort
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 0.02 mg/kg/Day | Cohort 2 0.08 mg/kg/Day | Cohort 3a 0.04 mg/kg/Day | Cohort 3b 0.06 mg/kg/Day | Total
Number analyzed (Participants) | 4 | 4 | 4 | 8 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.9 (2.9) | 10.2 (1.4) | 9.3 (1.4) | 11.2 (4.6) | 10.2 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 5 | 13
  Male | 2 | 1 | 1 | 3 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Aisan | 0 | 1 | 0 | 0 | 1
  Black | 0 | 0 | 0 | 1 | 1
  Caucasian | 4 | 3 | 4 | 7 | 18

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Profile of Omigapil:Maximum Observed Plasma Concentration (Cmax) of Omigapil
Time Frame: 0.5, 1, 1.5, 2, 4 and 8 hours post-dose on Day 1, Week 4 and Week 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Cohort 1 0.02 mg/kg/Day; Cohort 2 0.08 mg/kg/Day; Cohort 3a 0.04 mg/kg/Day; Cohort 3b 0.06 mg/kg/Day: Omigapil Treatment Oral Administration once per day after breakfast
Arm/Group | Cohort 1 0.02 mg/kg/Day | Cohort 2 0.08 mg/kg/Day | Cohort 3a 0.04 mg/kg/Day | Cohort 3b 0.06 mg/kg/Day
Number analyzed (Participants) | 4 | 4 | 4 | 8
ng/mL
  Day1 | 1.05 (32.4) | 4.75 (24.9) | 2.15 (62.8) | 3.27 (86.4)
  Week 4 | 1.10 (55.1) | 10.5 (57.3) | 1.98 (31.2) | 2.90 (96.1)
  Week 12 | 1.25 (37.8) | 11.6 (51.6) | 1.95 (31.9) | 3.43 (55.2)

2. Primary Outcome: Pharmacokinetic Profile of Omigapil: Time at Which Cmax Was Apparent (Tmax) of Omigapil
Time Frame: 0.5, 1, 1.5, 2, 4 and 8 hours post-dose on Day 1, Week 4 and Week 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Cohort 1 0.02 mg/kg/Day | Cohort 2 0.08 mg/kg/Day | Cohort 3a 0.04 mg/kg/Day | Cohort 3b 0.06 mg/kg/Day
Number analyzed (Participants) | 4 | 4 | 4 | 8
h
  Day 1 | 0.8 (3.9) | 0.8 (1.5) | 0.8 (3.9) | 0.5 (4.0)
  Week 4 | 0.6 (1.5) | 0.5 (2.0) | 0.5 (1.0) | 1.0 (4.0)
  Week 12 | 1.00 (1.6) | 0.9 (1.4) | 0.8 (1.0) | 1.0 (4.0)

3. Primary Outcome: Pharmacokinetic Profile of Omigapil Area Under the Plasma Concentration Versus Time Curve From Time Zero to 8h Post-dose (AUC0-8)
Time Frame: 0 to 8 hours post-dose on Day 1, Week 4, Week 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg.h/ml
Arm/Group | Cohort 1 0.02 mg/kg/Day | Cohort 2 0.08 mg/kg/Day | Cohort 3a 0.04 mg/kg/Day | Cohort 3b 0.06 mg/kg/Day
Number analyzed (Participants) | 4 | 4 | 4 | 8
mg.h/ml
  Day 1 | 3.37 (23.0) | 15.7 (38.5) | 7.12 (34.4) | 10.8 (69.5)
  Week 4 | 3.47 (48.2) | 29.7 (64.1) | 8.28 (15.7) | 11.0 (77.8)
  Week 12 | 3.79 (47.9) | 37.5 (31.0) | 6.91 (18.5) | 12.5 (91.6)

4. Secondary Outcome: Summary of All Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs reported during the treatment period
Time Frame: 12 weeks
Measure: Number; unit: number of events
Arm/Group | Cohort 1 0.02 mg/kg/Day | Cohort 2 0.08 mg/kg/Day | Cohort 3a 0.04 mg/kg/Day | Cohort 3b 0.06 mg/kg/Day
Number analyzed (Participants) | 4 | 4 | 4 | 8
number of events
  Treatment-emergent TEAEs | 41 | 40 | 29 | 75
  Serious TEAEs | 0 | 0 | 0 | 0
  Fatal TEAEs | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs (TEAEs) collected during the 12 weeks of treatment
Arm/Group | Cohort 1 0.02 mg/kg/Day | Cohort 2 0.08 mg/kg/Day | Cohort 3a 0.04 mg/kg/Day | Cohort 3b 0.06 mg/kg/Day
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/8
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 4/4 | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 0.02 mg/kg/Day (N=4) | Cohort 2 0.08 mg/kg/Day (N=4) | Cohort 3a 0.04 mg/kg/Day (N=4) | Cohort 3b 0.06 mg/kg/Day (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Faeces discoloured (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stoma site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Exposure to communicable disease (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Granulocyte count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Protein total decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary function test decreased (Investigations) | 2 (2) | 1 (1) | 3 (3) | 4 (5)
Red blood cells urine (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ultrasound liver abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cells urine positive (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (12)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Anorexia and bulimia syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Attention déficit / hyperactivity disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Ketonuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (3) | 3 (8) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 1 (3) | 4 (9) | 2 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Cooperative Research and Development Agreement

DOCUMENTS (2):
  • Study Protocol (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT01805024/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/24/NCT01805024/SAP_001.pdf